CLINICAL TRIAL: NCT06791642
Title: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique: a Multicenter Study of Clinical Outcomes, Recurrence Rates, and Quality of Life Improvements
Brief Title: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique:
Acronym: APOLLO
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, PhD, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 20252819
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Parastomal Hernia
Keywords: stoma; hernia; Laparoscopic repair
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Parietex™ Composite Mesh: Group 1: Parietex™ Composite Mesh
  This group consisted of patients who had their PSH repair performed using the Parietex™ Composite Mesh, a dual-layer synthetic mesh designed to promote tissue integration while minimizing the risk of adhesions. The Parietex™ mesh is composed of a macroporous structure on one side, which facilitates tissue ingrowth, and an anti-adhesive barrier on the other side to reduce complications such as bowel adhesions or erosion. This mesh was applied using the sandwich technique, combining a keyhole configuration around the stoma with an overlay reinforcement of the abdominal wall.
  Interventions: Device: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique
- Group 2: Synecor™ Hybrid Mesh: This group included patients who underwent PSH repair using the Synecor™ Hybrid Mesh, an advanced composite mesh that combines biologic and synthetic materials. The Synecor™ mesh integrates a bioresorbable layer for improved biocompatibility and tissue integration with a synthetic layer to enhance long-term strength and durability. It also incorporates anti-adhesive properties to minimize the risk of complications. Similar to the Parietex™ group, this mesh was used in the sandwich technique to provide dual-layer reinforcement.
  Key features of this group:
  * Mesh composition: Hybrid with bioresorbable and synthetic components for strength and tissue integration.
  * Clinical outcomes assessed: Recurrence rates, SSIs, seromas, and mesh-related complications, including hematomas or bulging.
  Interventions: Device: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique

INTERVENTIONS:
Device: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique — The sandwich technique was performed laparoscopically according to minimally invasive principles. Pneumoperitoneum was typically established using a Veress needle if the subcostal region was free from previous surgical scarring. For patients with prior extensive abdominal surgeries, a small laparotomy was performed to place the first 10-mm trocar directly under vision, ensuring safe entry into the peritoneal cavity. A 30° laparoscope was used throughout the procedure for enhanced visualization of the operative field.
  Trocar placement was designed to optimize access and ergonomics. The primary trocar was placed either in the periumbilical region or in the left or right flank, depending on the patient's anatomy and stoma location. Mesh used:1. Parietex™ Composite Mesh (Medtronic, USA): A multifilament polyester mesh with an anti-adhesive collagen barrier to minimize visceral adhesions.
  Groups: Group 1: Parietex™ Composite Mesh
Device: Laparoscopic Parastomal Hernia Repair Using the Sandwich Technique — The sandwich technique was performed laparoscopically according to minimally invasive principles. Pneumoperitoneum was typically established using a Veress needle if the subcostal region was free from previous surgical scarring. For patients with prior extensive abdominal surgeries, a small laparotomy was performed to place the first 10-mm trocar directly under vision, ensuring safe entry into the peritoneal cavity. A 30° laparoscope was used throughout the procedure for enhanced visualization of the operative field.
  Trocar placement was designed to optimize access and ergonomics. The primary trocar was placed either in the periumbilical region or in the left or right flank, depending on the patient's anatomy and stoma location. Mesh use Synecor™ Hybrid Mesh (BD, USA): A macroporous mesh combining polypropylene with a bioresorbable layer that degrades over time, leaving a durable support structure to promote tissue integration.
  Groups: Group 2: Synecor™ Hybrid Mesh

SUMMARY:
This study focuses on improving the surgical repair of parastomal hernias (PSHs), which are a common complication for patients with stomas. The investigators are examining the effectiveness of a specific technique called the "sandwich method," which uses two layers of mesh to reinforce the hernia site and reduce recurrence. The objective is to evaluate how well this method works over time, assess its impact on patient recovery and quality of life, and compare outcomes for different types of surgical materials used. This research aims to provide clearer guidance for surgeons and improve long-term results for patients undergoing PSH repair.

DETAILED DESCRIPTION:
Study Description: Improving Surgical Outcomes for Parastomal Hernia Repair

Parastomal hernias (PSHs) are a common and challenging complication that occurs in patients with stomas-surgically created openings in the abdomen used to divert waste. These hernias can cause discomfort, limit daily activities, and require surgical intervention to repair. Despite advancements in surgical techniques, PSH repair remains a complex issue, with high recurrence rates and varying outcomes.

This study investigates the effectiveness of a specific surgical approach called the "sandwich technique" for PSH repair. This method uses two layers of mesh to reinforce the abdominal wall and provide extra support around the stoma, aiming to reduce the likelihood of hernia recurrence while maintaining the function of the stoma. The first layer of mesh is placed directly around the stoma in a "keyhole" fashion, and the second layer reinforces the surrounding abdominal wall in a broader "overlay" configuration.

The research evaluates multiple aspects of this technique:

1. Effectiveness: Measuring recurrence rates over time, particularly for patients with larger hernias or recurrent hernias.
2. Safety: Assessing complications such as infections, seromas (fluid accumulation), or mesh-related issues.
3. Quality of Life (QoL): Using patient-reported surveys to evaluate how the repair impacts physical comfort, stoma care, body image, and social activities.
4. Comparison of Materials: Analyzing outcomes for two commonly used mesh types-Parietex™ Composite Mesh and Synecor™ Hybrid Mesh-to determine if material selection affects long-term results.

The study incorporates the European Hernia Society (EHS) classification system to categorize hernia types based on size and complexity. This allows for a tailored approach to treatment and helps identify which patients may benefit most from specific surgical strategies.

While the sandwich technique has shown promise in reducing recurrence rates and enhancing recovery, this research seeks to provide stronger evidence to guide surgeons in selecting the best techniques and materials for PSH repair. By focusing on patient-centered outcomes and refining surgical methods, the study aims to improve long-term results and overall quality of life for individuals living with stomas.

ELIGIBILITY:
Inclusion Criteria:

* Specify the criteria for participating in the study in a bulleted list under each category heading ("Inclusion Criteria" and "Exclusion Criteria"). Include only one item per bullet.

Exclusion Criteria:

Age below 18 years.

* Patients with recurrent parastomal hernia repairs requiring an open surgical approach.
* Evidence of active abdominal infection or sepsis at the time of surgery.
* Known allergies to mesh materials used in the study (e.g., Parietex™ or Synecor™).
* Presence of significant comorbidities making laparoscopic surgery unsafe (e.g., advanced cardiopulmonary disease).
* Pregnancy at the time of surgery.
* Inability to provide informed consent or comply with follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with a diagnosed parastomal hernia who are referred for surgical repair at participating hospitals. These patients are representative of individuals commonly managed in general and colorectal surgery practices, and they will be selected from both inpatient and outpatient settings.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
hernia recurrence rate | 12 months
  defined as clinical or radiological confirmation of a recurrent parastomal hernia.
hernia recurrence rate | 24 months
  defined as clinical or radiological confirmation of a recurrent parastomal hernia.

SECONDARY OUTCOMES:
Surgical Site Infections (SSIs) | 1 months
  The occurrence of surgical site infections was assessed as a critical indicator of postoperative morbidity. SSIs were monitored through clinical evaluations, including signs of redness, swelling, warmth, pain, and discharge at the surgical site, and were managed according to established guidelines.
Surgical Site Infections (SSIs) | 3 months
  The occurrence of surgical site infections was assessed as a critical indicator of postoperative morbidity. SSIs were monitored through clinical evaluations, including signs of redness, swelling, warmth, pain, and discharge at the surgical site, and were managed according to established guidelines.
Surgical Site Infections (SSIs) | 6 months
  The occurrence of surgical site infections was assessed as a critical indicator of postoperative morbidity. SSIs were monitored through clinical evaluations, including signs of redness, swelling, warmth, pain, and discharge at the surgical site, and were managed according to established guidelines.
Surgical Site Infections (SSIs) | 12 months
  The occurrence of surgical site infections was assessed as a critical indicator of postoperative morbidity. SSIs were monitored through clinical evaluations, including signs of redness, swelling, warmth, pain, and discharge at the surgical site, and were managed according to established guidelines.
Surgical Site Infections (SSIs) | 24 months
  The occurrence of surgical site infections was assessed as a critical indicator of postoperative morbidity. SSIs were monitored through clinical evaluations, including signs of redness, swelling, warmth, pain, and discharge at the surgical site, and were managed according to established guidelines.
Number of Participants with Postoperative Seroma Formation | 1 months
  Accumulation of fluid at the surgical site, confirmed through physical examination or imaging.
Number of Participants with Postoperative Seroma Formation: | 3 months
  Accumulation of fluid at the surgical site, confirmed through physical examination or imaging.
Number of Participants with Postoperative Seroma Formation: | 6 months
  Accumulation of fluid at the surgical site, confirmed through physical examination or imaging.
Number of Participants with Postoperative Seroma Formation: | 12 months
  Accumulation of fluid at the surgical site, confirmed through physical examination or imaging.
Number of Participants with Postoperative Seroma Formation: | 24 months
  Accumulation of fluid at the surgical site, confirmed through physical examination or imaging.
Number of Participants with Postoperative Hematoma Formation | 1 months
  Localized blood collection near the surgical site, evaluated clinically or with imaging as needed.
Number of Participants with Postoperative Hematoma Formation | 3 months
  Localized blood collection near the surgical site, evaluated clinically or with imaging as needed.
Number of Participants with Postoperative Hematoma Formation | 6 months
  Localized blood collection near the surgical site, evaluated clinically or with imaging as needed.
Number of Participants with Postoperative Hematoma Formation | 12 months
  Localized blood collection near the surgical site, evaluated clinically or with imaging as needed.
Number of Participants with Postoperative Hematoma Formation | 24 months
  Localized blood collection near the surgical site, evaluated clinically or with imaging as needed.
Mesh-Related Complications:Bowel Adhesions | until 24 months
  Abnormal fibrous connections between the bowel and mesh, potentially causing pain or obstruction.
Mesh-specific complications : Mesh Migration: | until 24 month
  Displacement of the mesh from its intended position.
Mesh-Related Complications:Mesh Erosion into the Stoma | until 24 months
  Displacement of the mesh from its intended position.
Number of Participants with Postoperative Bowel Obstruction | until 24 months
  Episodes of bowel obstruction were recorded based on patient symptoms (e.g., abdominal distension, vomiting) and confirmed using imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: francesco pizza, PhD, Study Director — Azienda Sanitaria Locale Napoli 2 Nord
Locations (1):
- francesco Pizza, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Explanation for Not Sharing Individual Participant Data (IPD)
  Individual participant data (IPD) will not be shared due to the following considerations:
  1. Patient Confidentiality: Sharing IPD may risk breaching participant privacy, even if anonymized, particularly given the detailed nature of surgical and clinical data.
  2. Ethical Constraints: The consent obtained from participants does not include provisions for data sharing beyond the scope of this study.
  3. Regulatory Compliance: Institutional policies and local regulations may limit the sharing of sensitive health information.
  4. Data Ownership: The data is collected across multiple centers, and permissions for sharing may vary depending on institutional agreements and data governance policies.
  5. Limited Generalizability of Raw Data: Given the study's small sample size and highly specialized focus, the broader utility of the raw IPD for external analysis is limited.

REFERENCES:
- [Background] Antoniou SA, Agresta F, Garcia Alamino JM, Berger D, Berrevoet F, Brandsma HT, Bury K, Conze J, Cuccurullo D, Dietz UA, Fortelny RH, Frei-Lanter C, Hansson B, Helgstrand F, Hotouras A, Janes A, Kroese LF, Lambrecht JR, Kyle-Leinhase I, Lopez-Cano M, Maggiori L, Mandala V, Miserez M, Montgomery A, Morales-Conde S, Prudhomme M, Rautio T, Smart N, Smietanski M, Szczepkowski M, Stabilini C, Muysoms FE. European Hernia Society guidelines on prevention and treatment of parastomal hernias. Hernia. 2018 Feb;22(1):183-198. doi: 10.1007/s10029-017-1697-5. Epub 2017 Nov 13. PMID 29134456